CLINICAL TRIAL: NCT05375682
Title: Integrating Care for Patients With Alcohol Liver Disease and Mental Health and Alcohol Use Disorders: A Pilot Study
Brief Title: Integrating Care for Patients With Alcohol Liver Disease and Alcohol Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Nabiha Faisal, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HS24921
Record Dates: First submitted 2022-05-03; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Alcohol; Liver
Keywords: Collaborative care; Integrated care; alcohol use disorder; Addiction medicine; cirrhosis; Alcohol liver disease; Alcoholic hepatitis
MeSH Terms: conditions — Liver Diseases, Alcoholic; Alcoholism; Fibrosis; Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated care program (Experimental): ICP intervention consists of several core intervention components.
  Interventions: Other: Integrated care program

INTERVENTIONS:
Other: Integrated care program — Core Component 1: Fostering Collaboration and Capacity Core Component 2: Streamlined communication process for referrals and care planning Core Component 3: Coordinated Care Conferences

SUMMARY:
Alcohol related liver disease (ALD) contributes to 50% cases of cirrhosis worldwide and is the leading indication for liver transplant in North America. The treatment for ALD is achieving total alcohol abstinence and preventing relapse as medical and surgical options are limited when drinking continues. Patient care has been hindered by the isolation of Addiction Medical Services from Internal Medicine, Family Medicine, and Hepatology. Patients with ALD would benefit from multidisciplinary approach as it combines medical care of liver disease and management of addiction and mental health. The investigators aim to develop a patient-centered integrated care pathway supported by expertise from Hepatology, Addiction Medicine and Psychiatry to improve access to addiction services for patients with ALD. By participating in the services, patients will experience decreased substance use, psychological symptoms, and improved health-related quality of life, with greater patient and provider satisfaction.

DETAILED DESCRIPTION:
Introduction: Alcohol Use Disorder (AUD) elevates the risk of a number of health conditions, with social, economic and clinical consequences. The effects of AUD are particular evident among individuals with ALD. The persistence of alcohol consumption is the main risk factor for progression of liver damage and complications. Despite this disease burden the resources devoted to either research or treatment of ALD have lagged compared with liver diseases from other etiologies. Progress has been hindered by the isolation of key specialites, which leads to late recognition of ALD. Patients with ALD would benefit from a multidisciplinary approach as it combines several domains including medical and psychiatric care; however, there is little research describing an integrated care alcohol use disorder (AUD) model for patients with ALD within Canada. Our multidisciplinary team, encompassing Hepatologists, Addiction Medicine and Psychiatry has been co-developing a patient-centered integrated care pathway to enhance collaborative practice among these specialities and meet the needs of our patients with ALD and AUD. The goal of this study is to carry out collaborative participatory research with health care providers and patients to co-develop and refine a responsive integrated care pathway (ICP) that addresses alcohol use disorders for patients with ALD at a large urban based hospital setting. Specifically, this study aims to:

1. To examine the feasibility of implementing several key strategies to initiate an integrated care pathway.
2. To explore the providers' and patients' perspectives regarding the acceptability of the integrated care pathway and seek their recommendations for improvement.
3. To explore the preliminary effects of the intervention based on changes over 6 months in health outcomes and use of health services.
4. To make recommendations that will inform spread and scale to other sites and for other conditions related to AUD.

Study design: This demonstration project will use a multi-method design to co-develop an integrated care pathway (ICP) for AUD and ALD, and to acquire the most comprehensive understanding of processes and outcomes. This will be a single site pragmatic pilot study evaluating feasibility, acceptability and preliminary effects of the ICP.

Participants: Investigators will use a convenience sample of consecutive ALD patients who are referred to the outpatient advanced liver clinic.

The intervention protocol: The 6-month ICP intervention consists of several core intervention components, building upon the available resources and usual care practices at Health Sciences Centre and based on an AUD/ALD model of care implemented elsewhere.

Data: Over the intervention period of the study, data on ICP implementation will be collected through monthly research team meetings with the interventionists, and through semi-structured interviews with patients and focus groups with health care providers. Multiple questionnaires and clinical data will be used to examine feasibility measures and preliminary clinical outcomes. Impact: The impact of this research is two-fold: 1) the combination of psychosocial interventions, pharmacological therapy and medical management offers the most effective strategy for addressing AUD among patients with ALD; 2) the collaboration and cooperation fostered through a participatory approach will tailor high quality care and enable our team to expand our model and develop community partnerships for spread and scale.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or biopsy-proven alcohol-associated cirrhosis or acute alcoholic hepatitis,
* Active drinking of any amount within the last 6 months,
* Willingness to speak with Addiction Medicine physicians

Exclusion Criteria:

* Not meeting all inclusion criteria
* Co-morbid severe mental illness
* Medically unstable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the ICP | One year
  Acceptability is a key element based on patients' and providers' perceptions/ experiences with the ICP and an overall evaluation of whether the intervention is agreeable and satisfactory. From patient participant interviews, conducted at the end of the study, investigators will explore perceptions and experiences in accessing and obtaining addiction service, perceived impact, benefit, and convenience. Investigators will conduct focus group discussions to seek health care providers' perspectives and experiences with AUD management challenges, the acceptability and use of the ICP, as well as where further support or improvements are needed.
Retention to the ICP | One year
  Retention will be determined with the (interventionist's) logs use to record visits with patients' and intervention uptake rates (use of pharmacotherapy, CBT/behavioral therapy, peer support group etc.).

SECONDARY OUTCOMES:
Change from baseline in the severity of alcohol use according to AUDIT (Alcohol Use Disorders Identification Test) score at 6 months after enrollment. | 6 months
  Minimum value: 0. Maximum value: 40. Higher scores indicate more severity of alcohol use.
Change from baseline in quality of life according to EQ-5D-5L questionnaire descriptive system (5-digit number that describes the patient's health state) at 6 months after enrollment. | 6 months
  The EQ-5D-5L (5-level EQ-5D version (EQ-5D-5L) by the EuroQol Group) (43) is a generic test to assess quality of life related to health. It includes 5 dimensions of quality of life (mobility, self-care, daily activities, pain, anxiety/depression) as a description of the patient's health state. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change from baseline in quality of life according to EQ-5D-5L questionnaire visual analogue scale (EQ VAS): patient's self-rated health from 0 to 100 at 6 months after enrollment. | 6 months
  The EQ-5D-5L (5-level EQ-5D version (EQ-5D-5L) by the EuroQol Group) is a generic test to assess quality of life related to health. It includes the EQ VAS, which records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled from score 100 ('The best health you can imagine') to 0 ('The worst health you can imagine'). The VAS can be used as a quantitative measure of health outcome.
Change in number of hospital admissions at 6 months after enrollment compared to previous six months. | One year
  Use of Health services
Change in number of Emergency Department Visits at 6 months after enrollment compared to previous six months. | One year
  Use of Health services

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolton JM, Leong C, Ekuma O, Prior HJ, Konrad G, Enns J, Singal D, Nepon J, Paille MT, Finlayson G, Nickel NC. Health service use among Manitobans with alcohol use disorder: a population-based matched cohort study. CMAJ Open. 2020 Nov 24;8(4):E762-E771. doi: 10.9778/cmajo.20200124. Print 2020 Oct-Dec. PMID 33234583
- [Background] Osna NA, Donohue TM Jr, Kharbanda KK. Alcoholic Liver Disease: Pathogenesis and Current Management. Alcohol Res. 2017;38(2):147-161. doi: 10.35946/arcr.v38.2.01. PMID 28988570
- [Background] Crabb DW, Im GY, Szabo G, Mellinger JL, Lucey MR. Diagnosis and Treatment of Alcohol-Associated Liver Diseases: 2019 Practice Guidance From the American Association for the Study of Liver Diseases. Hepatology. 2020 Jan;71(1):306-333. doi: 10.1002/hep.30866. No abstract available. PMID 31314133
- [Background] Grant BF, Chou SP, Saha TD, Pickering RP, Kerridge BT, Ruan WJ, Huang B, Jung J, Zhang H, Fan A, Hasin DS. Prevalence of 12-Month Alcohol Use, High-Risk Drinking, and DSM-IV Alcohol Use Disorder in the United States, 2001-2002 to 2012-2013: Results From the National Epidemiologic Survey on Alcohol and Related Conditions. JAMA Psychiatry. 2017 Sep 1;74(9):911-923. doi: 10.1001/jamapsychiatry.2017.2161. PMID 28793133
- [Background] Kanwal F, Kramer J, Asch SM, El-Serag H, Spiegel BM, Edmundowicz S, Sanyal AJ, Dominitz JA, McQuaid KR, Martin P, Keeffe EB, Friedman LS, Ho SB, Durazo F, Bacon BR. An explicit quality indicator set for measurement of quality of care in patients with cirrhosis. Clin Gastroenterol Hepatol. 2010 Aug;8(8):709-17. doi: 10.1016/j.cgh.2010.03.028. Epub 2010 Apr 10. PMID 20385251
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of alcohol-related liver disease. J Hepatol. 2018 Jul;69(1):154-181. doi: 10.1016/j.jhep.2018.03.018. Epub 2018 Apr 5. No abstract available. PMID 29628280
- [Background] Erim Y, Bottcher M, Schieber K, Lindner M, Klein C, Paul A, Beckebaum S, Mayr A, Helander A. Feasibility and Acceptability of an Alcohol Addiction Therapy Integrated in a Transplant Center for Patients Awaiting Liver Transplantation. Alcohol Alcohol. 2016 Jan;51(1):40-6. doi: 10.1093/alcalc/agv075. Epub 2015 Jun 28. PMID 26124208
- [Background] Mellinger JL, Winder GS, Fernandez AC, Klevering K, Johnson A, Asefah H, Figueroa M, Buchanan J, Blow F, Lok ASF. Feasibility and early experience of a novel multidisciplinary alcohol-associated liver disease clinic. J Subst Abuse Treat. 2021 Nov;130:108396. doi: 10.1016/j.jsat.2021.108396. Epub 2021 Apr 9. PMID 34118717
- [Background] Winder GS, Fernandez AC, Klevering K, Mellinger JL. Confronting the Crisis of Comorbid Alcohol Use Disorder and Alcohol-Related Liver Disease With a Novel Multidisciplinary Clinic. Psychosomatics. 2020 May-Jun;61(3):238-253. doi: 10.1016/j.psym.2019.12.004. Epub 2019 Dec 19. PMID 32033835
- [Background] Rehm J, Mathers C, Popova S, Thavorncharoensap M, Teerawattananon Y, Patra J. Global burden of disease and injury and economic cost attributable to alcohol use and alcohol-use disorders. Lancet. 2009 Jun 27;373(9682):2223-33. doi: 10.1016/S0140-6736(09)60746-7. PMID 19560604
- [Background] Hulme J, Sheikh H, Xie E, Gatov E, Nagamuthu C, Kurdyak P. Mortality among patients with frequent emergency department use for alcohol-related reasons in Ontario: a population-based cohort study. CMAJ. 2020 Nov 23;192(47):E1522-E1531. doi: 10.1503/cmaj.191730. PMID 33229348
- [Background] Hobin E, Smith B. Is another public health crisis brewing beneath the COVID-19 pandemic? Can J Public Health. 2020 Jun;111(3):392-396. doi: 10.17269/s41997-020-00360-z. Epub 2020 Jun 18. PMID 32557350
- [Background] Pollard MS, Tucker JS, Green HD Jr. Changes in Adult Alcohol Use and Consequences During the COVID-19 Pandemic in the US. JAMA Netw Open. 2020 Sep 1;3(9):e2022942. doi: 10.1001/jamanetworkopen.2020.22942. PMID 32990735
- [Background] Beste LA, Harp BK, Blais RK, Evans GA, Zickmund SL. Primary Care Providers Report Challenges to Cirrhosis Management and Specialty Care Coordination. Dig Dis Sci. 2015 Sep;60(9):2628-35. doi: 10.1007/s10620-015-3592-1. Epub 2015 Mar 3. PMID 25732712
- [Background] Grant BF, Goldstein RB, Saha TD, Chou SP, Jung J, Zhang H, Pickering RP, Ruan WJ, Smith SM, Huang B, Hasin DS. Epidemiology of DSM-5 Alcohol Use Disorder: Results From the National Epidemiologic Survey on Alcohol and Related Conditions III. JAMA Psychiatry. 2015 Aug;72(8):757-66. doi: 10.1001/jamapsychiatry.2015.0584. PMID 26039070
- [Background] Mellinger JL, Fernandez A, Shedden K, Winder GS, Fontana RJ, Volk ML, Blow FC, Lok ASF. Gender Disparities in Alcohol Use Disorder Treatment Among Privately Insured Patients with Alcohol-Associated Cirrhosis. Alcohol Clin Exp Res. 2019 Feb;43(2):334-341. doi: 10.1111/acer.13944. Epub 2019 Jan 22. PMID 30667521
- [Background] Mellinger JL, Scott Winder G, DeJonckheere M, Fontana RJ, Volk ML, Lok ASF, Blow FC. Misconceptions, preferences and barriers to alcohol use disorder treatment in alcohol-related cirrhosis. J Subst Abuse Treat. 2018 Aug;91:20-27. doi: 10.1016/j.jsat.2018.05.003. Epub 2018 May 18. PMID 29910011
- [Background] Bradley KA, Kivlahan DR. Bringing patient-centered care to patients with alcohol use disorders. JAMA. 2014 May 14;311(18):1861-2. doi: 10.1001/jama.2014.3629. No abstract available. PMID 24825640
- [Background] Goodwin N. Understanding Integrated Care. Int J Integr Care. 2016 Oct 28;16(4):6. doi: 10.5334/ijic.2530. No abstract available. PMID 28316546
- [Background] Moffat K, Mercer SW. Challenges of managing people with multimorbidity in today's healthcare systems. BMC Fam Pract. 2015 Oct 14;16:129. doi: 10.1186/s12875-015-0344-4. PMID 26462820
- [Background] Donald M, Dower J, Kavanagh D. Integrated versus non-integrated management and care for clients with co-occurring mental health and substance use disorders: a qualitative systematic review of randomised controlled trials. Soc Sci Med. 2005 Mar;60(6):1371-83. doi: 10.1016/j.socscimed.2004.06.052. PMID 15626531
- [Background] O'Toole TP, Strain EC, Wand G, McCaul ME, Barnhart M. Outpatient treatment entry and health care utilization after a combined medical/substance abuse intervention for hospitalized medical patients. J Gen Intern Med. 2002 May;17(5):334-40. doi: 10.1046/j.1525-1497.2002.10638.x. PMID 12047729
- [Background] Weisner C, Mertens J, Parthasarathy S, Moore C, Lu Y. Integrating primary medical care with addiction treatment: a randomized controlled trial. JAMA. 2001 Oct 10;286(14):1715-23. doi: 10.1001/jama.286.14.1715. PMID 11594896
- [Background] Saxon AJ, Malte CA, Sloan KL, Baer JS, Calsyn DA, Nichol P, Chapko MK, Kivlahan DR. Randomized trial of onsite versus referral primary medical care for veterans in addictions treatment. Med Care. 2006 Apr;44(4):334-42. doi: 10.1097/01.mlr.0000204052.95507.5c. PMID 16565634
- [Background] Reus VI, Fochtmann LJ, Bukstein O, Eyler AE, Hilty DM, Horvitz-Lennon M, Mahoney J, Pasic J, Weaver M, Wills CD, McIntyre J, Kidd J, Yager J, Hong SH. The American Psychiatric Association Practice Guideline for the Pharmacological Treatment of Patients With Alcohol Use Disorder. Focus (Am Psychiatr Publ). 2019 Apr;17(2):158-162. doi: 10.1176/appi.focus.17205. Epub 2019 Apr 10. PMID 32021585
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Weinrieb RM, Van Horn DH, Lynch KG, Lucey MR. A randomized, controlled study of treatment for alcohol dependence in patients awaiting liver transplantation. Liver Transpl. 2011 May;17(5):539-47. doi: 10.1002/lt.22259. PMID 21506242
- [Background] Johnson JA, Coons SJ. Comparison of the EQ-5D and SF-12 in an adult US sample. Qual Life Res. 1998 Feb;7(2):155-66. doi: 10.1023/a:1008809610703. PMID 9523497